CLINICAL TRIAL: NCT07253961
Title: The Effects of Lateral Neck Cold Application for Vagal Nerve Stimulation on Pain During Peripheral Venous Cannulation in Obese Patients: A Prospective Randomized Controlled Study
Brief Title: Cold-Induced Vagal Stimulation for Attenuating Venipuncture Pain in Obese Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: venöz istinye
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Venipuncture Pain; Vagal Nerve Stimulation; Cold Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Application Group (Experimental): Participants will receive cold stimulation to the lateral neck region (over the sternocleidomastoid muscle) using a marble stone cooled to 0-4°C for 5 seconds immediately before peripheral venous cannulation.
  Interventions: Procedure: Cold Application to Lateral Neck Region
- Standard Venous Cannulation Group (Placebo Comparator): Participants will undergo routine peripheral venous cannulation without any prior intervention.
  Interventions: Procedure: Cold Application to Lateral Neck Region

INTERVENTIONS:
Procedure: Cold Application to Lateral Neck Region — Application of a marble stone cooled to 0-4°C on the lateral neck (over the sternocleidomastoid muscle) for 5 seconds prior to venous cannulation to stimulate the vagus nerve.

SUMMARY:
This prospective, randomized controlled clinical trial aims to evaluate the effect of lateral neck cold application for vagal nerve stimulation on pain perception during peripheral venous cannulation in obese patients. Venous cannulation is a routine but painful procedure, especially in individuals with a body mass index (BMI) greater than 30, who often have heightened pain sensitivity due to chronic inflammation.

Participants will be randomly assigned to one of two groups:

Group 1 (Cold Application Group): A cold marble stone (0-4°C) will be applied to the lateral neck region (over the sternocleidomastoid muscle) for 5 seconds immediately before venous cannulation.

Group 2 (Control Group): Standard venous cannulation will be performed without any prior intervention.

Pain intensity will be assessed using the Visual Analog Scale (VAS) immediately after cannulation. Hemodynamic parameters (heart rate, blood pressure, oxygen saturation, respiratory rate) will be recorded before and after the procedure.

The primary outcome is the difference in VAS scores between the two groups. Secondary outcomes include changes in hemodynamic parameters. The study will enroll 150 participants over approximately two months following ethics approval.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-72 years
* physical status I-III
* Scheduled for elective surgery
* Body Mass Index (BMI) > 30 kg/m²
* Provided written informed consent

Exclusion Criteria:

* Emergency surgical cases
* Oncologic surgery
* Pregnant patients
* History of hand dorsum surgery or scarring
* Psoriasis or other local skin lesions/infections at cannulation site
* Peripheral vascular disease
* Chronic analgesic, opioid, steroid, or gabapentinoid use
* Substance abuse history
* Peripheral neuropathy
* Previous or ongoing oncologic treatment
* Severe mental retardation or communication impairment preventing cooperation

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Venous cannulation pain (VAS, 0-10) | Immediately after cannulation (within ~1 minute)
  Pain intensity will be assessed once, right after peripheral venous cannulation, using a 10-cm Visual Analog Scale (0 = no pain, 10 = worst imaginable pain). The score will be recorded as a continuous variable and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Background] Jungmann M, Vencatachellum S, Van Ryckeghem D, Vogele C. Effects of Cold Stimulation on Cardiac-Vagal Activation in Healthy Participants: Randomized Controlled Trial. JMIR Form Res. 2018 Oct 9;2(2):e10257. doi: 10.2196/10257. PMID 30684416
- [Result] Agarwal A, Sinha PK, Tandon M, Dhiraaj S, Singh U. Evaluating the efficacy of the valsalva maneuver on venous cannulation pain: a prospective, randomized study. Anesth Analg. 2005 Oct;101(4):1230-1232. doi: 10.1213/01.ane.0000167270.15047.49. PMID 16192551
- [Result] Kumar S, Gautam SK, Gupta D, Agarwal A, Dhirraj S, Khuba S. The effect of Valsalva maneuver in attenuating skin puncture pain during spinal anesthesia: a randomized controlled trial. Korean J Anesthesiol. 2016 Feb;69(1):27-31. doi: 10.4097/kjae.2016.69.1.27. Epub 2016 Jan 28. PMID 26885298